CLINICAL TRIAL: NCT05416190
Title: Effect of Injectable Anticoagulants on Research for a Circulating Lupus-type Anticoagulant
Acronym: ANTICOLA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Clermont-Ferrand (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: AOI 2021 TALON; 2021-A02743-38 (Other: ANSM)
Record Dates: First submitted 2022-05-12; First posted 2022-06-13 (Actual); Last update posted 2024-06-21 (Actual); Status verified 2022-06

CONDITIONS: Antiphospholipid Syndrome; Anticoagulant Drugs
Keywords: Lupus coagulation inhibitor; Anticoagulant drugs
MeSH Terms: conditions — Antiphospholipid Syndrome

STUDY DESIGN:
Intervention Model Description: Citrated whole blood was collected from all participants and lupus anticoagulant testing was performed before and after spiking in vitro injectable anticoagulants. No distinction between the groups LA+ and LA-.
Masking Description: Patients are recruited according to their LA status (LA- or LA+).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group/Cohort 1 : (Other): Notion of the presence of lupus anticoagulant (according to ISTH criteria) and whose last test was positive
  Interventions: Diagnostic Test: Lupus anticoagulant testing
- Group/Cohort 2: (Other): Without a previous thrombosis and considered healthy on the basis of the interview and clinical examination. Without coagulation disease.
  Interventions: Diagnostic Test: Lupus anticoagulant testing

INTERVENTIONS:
Diagnostic Test: Lupus anticoagulant testing — The patient will have a visit during which a blood sample will be taken, a clinical examination will be performed, and data will be collected.

SUMMARY:
The aim is to assess the effect of injectable anticoagulants (unfractionated heparin (UFH), low molecular weight heparins (LMWH), fondaparinux, danaparoid, argatroban) on lupus anticoagulant testing assays over broad anti-Xa activity ranges and to establish their potential for causing false-positive or false-negative results.

DETAILED DESCRIPTION:
Citrated whole blood was collected from subjects with positive lupus anticoagulant (LA) testing and from subjects with negative LA testing. Injectable anticoagulants were prepared in demineralized water and added to plasma samples LA+ and LA- to obtain broad anti-Xa activity ranges. Anti-Xa measurement and LA testing were performed in neat and spiked plasma samples. LA testing was performed with 4 different analyzer-reagent combinations to represent almost all hemostasis manufacturers currently available. There will be no direct comparison between the LA+ and LA- groups, the objective is to evaluate the effect of increasing concentrations of injectable anticoagulants on these 2 distinct populations.

ELIGIBILITY:
Inclusion Criteria:

* For all subjects:
* Adult male or female subject.
* In capacity to give informed consent to participate in the research.
* Affiliated to a Social Security system.

For the LA- group:

* Without a previous thrombosis and considered healthy on the basis of the interview and clinical examination.
* Without coagulation disease

For the LA+ group:

- Notion of the presence of lupus anticoagulant (according to ISTH criteria) and whose last test was positive.

Exclusion Criteria:

For all subjects:

* Medical history considered by the investigator to be incompatible with the trial
* Refused participation
* Recent administration of oral or injectable anticoagulants
* INR > 1.5
* Pregnant women, nursing mothers
* Guardianship, curatorship, deprived of liberty, safeguard of justice

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 188 (Actual)
Dates: Start 2022-06-02 (Actual); Primary Completion 2024-05-21 (Actual); Study Completion 2024-05-21 (Actual)

PRIMARY OUTCOMES:
Results of lupus anticoagulant testing: positive or negative | day 1
  Concerning the impact of injectable anticoagulants on the final diagnosis of LA testing (negative or positive), in a population of LA+ and LA- subjects, particular attention will be paid to the study of false negatives and false positives expressed in % and 95% confidence intervals.

SECONDARY OUTCOMES:
Effect of injectable anticoagulants on the clotting times of each of the tests involved in LA testing (detection, mixing and confirmation tests). | day 1
  comparison of clotting times in the absence and presence of increasing concentrations of anticoagulants will be carried out by Anova or non-parametric Kruskal-Wallis test if the conditions of Anova are not respected. Graphical representations will be associated with these analyses.
Determination of the threshold limits of injectable anticoagulants (anti-Xa activities) allowing a reliable LA diagnosis, for each analytical solution tested (analyzer/reagent combinations). | day1
  comparison of clotting times in the absence and presence of increasing concentrations of anticoagulants will be carried out by Anova or non-parametric Kruskal-Wallis test if the conditions of Anova are not respected.

CONTACTS AND LOCATIONS:
Overall Officials: Laurie TALON, Principal Investigator — University Hospital, Clermont-Ferrand
Locations (1):
- CHU clermont-ferrand, Clermont-Ferrand, France